CLINICAL TRIAL: NCT01221779
Title: Chronic Aphasia - Improved by Intensive Training and Electrical Brain
Brief Title: Chronic Aphasia - Improved by Intensive Training and Electrical Brain Stimulation
Acronym: CATS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Marcus Meinzer, Creutzfeldt Fellow, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CATS01EO0801
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Post-Stroke Chronic Aphasia; Anomia (Word-retrieval Impairment)
Keywords: Intensive language therapy; Anomia; Magnetic Resonance Imaging
MeSH Terms: conditions — Anomia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham tDCS (Placebo Comparator)
  Interventions: Behavioral: Intensive language therapy
- anodal tDCS (Experimental)
  Interventions: Behavioral: Intensive language therapy

INTERVENTIONS:
Behavioral: Intensive language therapy — 2 weeks of daily computerized naming training, daily, 3 hours
  Arms: sham tDCS
Behavioral: Intensive language therapy — 2 weeks of daily computerized naming training, daily, 3 hours
  Arms: anodal tDCS

SUMMARY:
The purpose of this study is to determine if non-invasive electrical brain stimulation can enhance the out of intensive language therapy in chronic aphasia

DETAILED DESCRIPTION:
Stroke is the leading cause of death and disability worldwide. Given the increasing average lifespan worldwide, the incidence and prevalence of patients with stroke will dramatically increase in the future. One of the most frequent and devastating conditions after stroke is aphasia, which affects language production and comprehension. High-frequent intensive speech-and-language therapy is currently the treatment of choice in chronic aphasia. However, despite its general effectiveness, treatment effect sizes are only low to moderate. Thus, there is a pressing need to explore novel training-adjuvant therapies to enhance treatment efficacy. Moreover, very little is known about the neurobiology of treatment-induced recovery in chronic aphasia. This is the prerequisite to improve existing and/or develop new treatment paradigms.

Thus, in the present project we aim to assess whether the outcome of intensive language training can be enhanced by adjuvant non-invasive brain stimulation. We will be using anodal transcranial direct current stimulation (atDCS) that has previously been shown to enhance (a) language and motor learning in healthy subjects and (b) motor recovery in stroke patients. Specifically, in a longitudinal group comparison design, two matched groups of patients with chronic anomia will receive two weeks of intensive language training with or without atDCS. Treatment effects will be assessed immediately after the two week intervention period and several months after the end of the training. We will also use functional and structural magnetic resonance imaging (MRI) to elucidate language network changes in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* right-handedness
* single first time left-hemisphere stroke
* fluent- or non-fluent chronic aphasia (more than six months post-stroke)
* anomia (PR>10 and PR<60 Aachen Aphasia Naming Subtest)
* native German Speaker

Exclusion Criteria:

* more than one stroke
* alcoholism, severe psychiatric conditions, other neurological conditions
* other non-treated medical problems, severe microangiopathy
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Boston Naming Test | Change of naming score from baseline (day 1 of study) to immediately after 2-week intervention period (post-testing)

SECONDARY OUTCOMES:
Boston Naming Test | Change of naming score from post-testing (after end of intervention) to 3 months after the intervention (follow-up)
  The follow-up will be administered to assess the stability of the treatment gains
Naming performance during functional magnetic resonance scanning | Change of naming score from baseline (day 1 of study) to immediately after 2-week intervention period (post-testing)
  assessed during overt picture naming task
Naming performance during functional magnetic resonance imaging | Change of naming score from post-testing (after end of intervention) to 3 months after the intervention (follow-up)
  assessed during overt picture naming task

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Meinzer, PhD, Principal Investigator — Charite, University Medicine, Neurology; Agnes Flöel, MD, Study Director — Charite, University Medicine, Neurology
Locations (1):
- Charite, University Medicine, Dept. of Neurology, Berlin, Germany